CLINICAL TRIAL: NCT00615251
Title: A Phase 3, Single-Blind, Randomized Study to Compare DR-2011 to a Progesterone Gel for Luteal Phase Supplementation for In Vitro Fertilization
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of DR-2011 for In Vitro Fertilization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DR-PGN-302
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-08

CONDITIONS: Infertility
Keywords: In vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: DR-2011
- 2 (Active Comparator)
  Interventions: Drug: Crinone 8%

INTERVENTIONS:
Drug: DR-2011 — Progesterone vaginal ring for approximately 10 weeks
  Arms: 1
Drug: Crinone 8% — progesterone vaginal gel for approximately 10 weeks
  Arms: 2

SUMMARY:
This is a multi-center study to evaluate the effects of DR-2011 compared to a progesterone gel in women undergoing in vitro fertilization with fresh eggs. The overall study duration will be approximately 12 months and will involve ovarian suppression/stimulation protocols as well as egg retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal, aged 18-42 old at time of consent
* At least one cycle without fertility medication prior to screening
* Tubal, idiopathic, male factor, ovulatory dysfunction or endometriosis- linked infertility
* Semen analysis (frozen sperm, including donor sperm, may be used, as long as testing done at time of freezing meets standard criteria)
* Others as indicated by FDA-approved protocol

Exclusion Criteria:

* Any contraindication to progesterone therapy
* BMI > 38 kg/m2
* Clinically significant gynecologic pathology (for example: submucosal fibroids, abnormal uterine cavity, or others)
* History of more than 1 failed fresh IVF cycles
* More than 2 consecutive clinical miscarriages (gestational sac observed on ultrasound)
* Others as indicated by FDA-approved protocol

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1297 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate at 8 weeks and 12 weeks of pregnancy | 8 weeks of pregnancy (6 weeks after egg retrieval) and 12 weeks of pregnancy (10 weeks after egg retrieval)

SECONDARY OUTCOMES:
Secondary outcome measures will include: live birth rate, cycle cancellation rate, rate of spontaneous abortion, rate of biochemical pregnancy, rate of ectopic pregnancy | Duration of study
Adverse events | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Research Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (29):
- United States (29):
  - Duramed Investigational Site, Tarzana, California
  - Duramed Investigational Site, West Los Angeles, California
  - Duramed Investigational Site, Westlake, California
  - Duramed Investigational Site, Clearwater, Florida
  - Duramed Investigational Site, Alpharetta, Georgia
  - Duramed Investigational Site, Atlanta, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Chicago, Illinois
  - Duramed Investigational Site, Highland Park, Illinois
  - Duramed Investigational Site, Rockville, Maryland
  - Duramed Investigational Site, Dearborn, Michigan
  - Duramed Investigational Site, Flint, Michigan
  - Duramed Investigational Site, Rochester Hills, Michigan
  - Duramed Investigational Site, Saginaw, Michigan
  - Duramed Investigational Site, Ypsilanti, Michigan
  - Duramed Investigational Site, Woodbury, Minnesota
  - Duramed Investigational Site, Reno, Nevada
  - Duramed Investigational Site, Marlton, New Jersey
  - Duramed Investigational Site, Morristown, New Jersey
  - Duramed Investigational Site, Cincinnati, Ohio
  - Duramed Investigational Site, Sylvania, Ohio
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Mt. Pleasant, South Carolina
  - Duramed Investigational Site, Myrtle Beach, South Carolina
  - Duramed Investigational Site, Austin, Texas
  - Duramed Investigational Site, Beaumont, Texas
  - Duramed Investigational Site, Bedford, Texas
  - Duramed Investigational Site, Webster, Texas
  - Duramed Investigational Site, Norfolk, Virginia

REFERENCES:
- [Derived] Ginsburg ES, Jellerette-Nolan T, Daftary G, Du Y, Silverberg KM. Patient experience in a randomized trial of a weekly progesterone vaginal ring versus a daily progesterone gel for luteal support after in vitro fertilization. Fertil Steril. 2018 Nov;110(6):1101-1108.e3. doi: 10.1016/j.fertnstert.2018.07.014. PMID 30396554
- [Derived] Stadtmauer L, Silverberg KM, Ginsburg ES, Weiss H, Howard B. Progesterone vaginal ring versus vaginal gel for luteal support with in vitro fertilization: a randomized comparative study. Fertil Steril. 2013 May;99(6):1543-9. doi: 10.1016/j.fertnstert.2012.12.052. Epub 2013 Mar 4. PMID 23465817